CLINICAL TRIAL: NCT02715765
Title: The Use of Transcranial Electrical Stimulation for Hallucinations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left university, the grant could not be transferred, no data was collected
Sponsor: University of Minnesota (Other)
Collaborators: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSYCH-2016-24233
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham (Sham Comparator): The sham procedure involves only 40 sec direct current stimulation at 2mA and then drops to 0mA with 15msec pulses every 550msec.
  Interventions: Device: Transcranial Sham Stimulation
- Active tDCS (Experimental): Current (2mA) is initiated in a ramp-like fashion over 10s from 0mA to 2mA using (SPONSTIM-25 25cm2 electrodes). The current is held constant for 20 min. Then the current is decreased in a ramp-like fashion over 10s from 2mA to 0mA.
  Interventions: Device: Transcranial Direct Current Stimulation
- Active tRNS (Experimental): Current (2mA) is initiated in a ramp-like fashion over 10s from 0mA to 2mA using (SPONSTIM-25 25cm2 electrodes). Once at 2mA, an alternating current of 2mA with a 0mA offset is applied at random frequencies over a range of 0.1 to 100 Hz. This is performed for 20 minutes. Then the current is decreased in a ramp-like fashion over 10s from 2mA to 0mA.
  Interventions: Device: Transcranial Random Noise Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Energetic parameters are 2mA for 20 min with SPONSTIM-25 25cm2 electrodes. Current delivery is initiated in a ramp-like fashion over 10s from 0mA to 2mA. Once at 2mA, the current is held constant for the entire session. At the end of stimulation, current is decreased in a ramp-like fashion over 10s from 2mA to 0mA. Should the participant not be able to tolerate a current of 2mA due to pain or irritation, the current will be decreased down to a minimum of 1.5mA. If 1.5 mA is still not tolerable, the participant will be removed from the study. Electrode placement is based on the international 10-20 electrode placement system. The anode is placed at the midpoint between F3 and FP1, a location corresponding approximately to the left dorsolateral prefrontal cortex, and the cathode placed at the midpoint between T3 and P3, a location corresponding to left temporo-parietal junction
  Other Names: tdcs
  Arms: Active tDCS
Device: Transcranial Random Noise Stimulation — Energetic parameters are 2mA for 20 min with SPONSTIM-25 25cm2 electrodes. Current delivery is initiated in a ramp-like fashion over 10s from 0mA to 2mA. Once at 2mA, the current alternates at 2mA with a 0mA offset applied at random frequencies over a range of 0.1 to 100 Hz. At the end of stimulation, current is decreased in a ramp-like fashion over 10s from 2mA to 0mA. Should the participant not be able to tolerate a current of 2mA due to pain or irritation, the current will be decreased down to a minimum of 1.5mA. If 1.5 mA is still not tolerable, the participant will be removed from the study. Electrode placement is based on the international 10-20 electrode placement system. The anode is placed at the midpoint between F3 and FP1, a location corresponding approximately to the left dorsolateral prefrontal cortex, and the cathode placed at the midpoint between T3 and P3, a location corresponding to left temporo-parietal junction
  Other Names: trns
  Arms: Active tRNS
Device: Transcranial Sham Stimulation — Energetic parameters are 2mA for 20 min with SPONSTIM-25 25cm2 electrodes. The sham procedure involves only 40 sec stimulation at 2mA and then drops to 0mA with 15msec pulses every 550msec. Should the participant not be able to tolerate a current of 2mA due to pain or irritation, the current will be decreased down to a minimum of 1.5mA. If 1.5 mA is still not tolerable, the participant will be removed from the study. Electrode placement is based on the international 10-20 electrode placement system. The anode is placed at the midpoint between F3 and FP1, a location corresponding approximately to the left dorsolateral prefrontal cortex, and the cathode placed at the midpoint between T3 and P3, a location corresponding to left temporo-parietal junction
  Other Names: sham
  Arms: Sham

SUMMARY:
Schizophrenia is a serious mental health disorder that affects approximately 1% of the population. Auditory hallucinations are present in as many as 50-75% of patients with this diagnosis. The hallucinations experienced by patients vary greatly and can severely impact an individual's ability to function on a daily basis. In approximately 25-30% of these patients, medication is an ineffective mechanism for managing these symptoms. These hallucinations are known as medication refractory auditory hallucination (MRAH). For those whose auditory hallucinations do not respond to medication, non-surgical brain stimulation (NBS) has recently shown promise as a therapeutic intervention. Two specific types of NBS, called transcranial direct current stimulation (tDCS) and transcranial random noise stimulation (tRNS), seem particularly well suited to treating MRAH. They have yet to be compared to each other in large samples of patients with MRAH. The goal of the study is to investigate whether tRNS and tDCS are effective in the treatment of MRAH and if one is better than the other when compared directly.

DETAILED DESCRIPTION:
Purpose and Background

Schizophrenia is a serious mental health disorder with a constellation of positive, negative, and cognitive symptoms. Negative symptoms can include characteristics such as affective flattening, avolition, and alogia. Positive symptoms can include delusions, hallucinations, and disorganized speech or behavior. Auditory hallucinations (AH) are a hallmark of schizophrenia. They are reported in as many as 50-75% of patients with this diagnosis. The hallucinations experienced by patients vary greatly and can severely impact an individual's ability to function on a daily basis. In approximately 25-30% of patients diagnosed with schizophrenia, medication is an ineffective mechanism for managing these symptoms. These hallucinations are known as medication refractory auditory hallucinations (MRAH). They are defined as "the persistence of daily hallucinations without remission despite antipsychotic medication at an adequate dosage for at least three months".

For those whose AH do not respond to medication, non-surgical brain stimulation (NBS) has recently shown promise as a therapeutic intervention. Specifically, the use of conductive electrical approaches termed transcranial electrical stimulation (tES). One method of tES that has received renewed interest due to its high portability, safety, and modulatory effects is transcranial direct current stimulation (tDCS). tDCS involves applying a weak electrical current using saline soaked electrode sponges, causing either increases or decreases in cortical excitability, respectively. Research has shown in both healthy subjects and patients (e.g. Alzheimer's disease, Parkinson's disease, stroke, and depression) that tDCS has the potential to modulate synaptic and neurotransmitter-dependent plasticity underlying changes in behavior and learning. Brunelin et al utilized tDCS to successfully reduce MRAH in a population diagnosed with schizophrenia. They were able to reduce AH by approximately 30% in their sample after 5 days of twice-daily treatment and this effect was maintained for approximately three months following treatment. This finding has yet to be replicated in a similar study.

Along with tDCS, other new methods of NBS are being investigated across various disease states. One such study looked at the impact of tES on tinnitus. They tested whether type of tES made a difference in efficacy. They compared tDCS to tRNS. tRNS is very similar to tDCS except that it superimposes a random "white noise" gaussian waveform (from 0.1 hz to 640 hz) on top of the DC current. They found that tRNS induced a larger suppressive effect on tinnitus loudness and tinnitus-related distress when compared to tDCS. While their findings were in tinnitus, there are now multiple scholarly works describing a relationship of tinnitus and AH, possibly as a continuum or dimension underlying a variety of normal and disease states. This relationship suggests strategies found to be efficacious for tinnitus may in fact also be efficacious for AH. Recently, there was a case series showing possible efficacy in AH using tRNS.

The purpose of the study is to examine the efficacy of tES in the treatment of MRAH of schizophrenia. The hypothesis is that tRNS will provide a larger reduction of AH in those with schizophrenia as compared to tDCS and no treatment (i.e. sham). Confirmation of this hypothesis would provide an exciting new option for treatment and may provide an even higher level of efficacy than is seen in tDCS. Further, this study would also provide replication of the work by Brunelin et al. and further support of tES as a compelling tool for the management of severe MRAH.

Specific Aims

1. Determine efficacy of tES as a treatment for MRAH. Hypothesis 1a: tDCS is more effective than sham in the treatment of MRAH shown by a reduction in both total and subscores of the AHRS. Hypothesis 1b: tRNS is more effective than both sham and tDCS in the treatment of MRAH as shown by a reduction in both total and subscores of the AHRS.
2. Demonstrate safety and tolerability of tES in the treatment of MRAH. Hypothesis 2a: tDCS is safe and well tolerated in the treatment of MRAH as demonstrated by the TSEQ. Hypothesis 2a: tRNS is safe and well tolerated in the treatment of MRAH as demonstrated by TSEQ.
3. Exploratory: Detect tES sensitive subtypes of AH based on the MUPS.

Study Design

This study is double-blind, between group, and sham-controlled. Subjects will be randomized to one of three arms (tRNS, tDCS, or sham) and will remain in that arm for the duration of the study. All subjects will complete an enrollment visit, ten treatment visits (2 visits per day), and 1, 3, and 6 month follow-up visits. Given that durability of effect has been suggested in the literature to be less than 6 months, patients will not be followed beyond 6 months. The outcome of this study will be measured by standard auditory hallucination rating scales including the Positive and Negative Symptoms Scale (PANSS), Auditory Hallucinations Rating Scale (AHRS), and psychotic symptom rating scales (PSYRATS). Both the AHRS and PSYRATS are included as outcome measures to ensure generalizability to existing studies on tES (which use the AHRS) along with the broader body of AH research (which use the PSYRATS). The primary efficacy parameter will be the PSYRATS as this has shown the most evidence for accurate representation of AH.

Clinical Significance

* This study will replicate and expand on previous research regarding the use of tES as a treatment for medication refractory auditory hallucinations
* Based on the findings, this study could have potential application as a non-invasive clinical intervention for treating MRAH which affect 25% of medicated patients with schizophrenia.

Subjects

This study will recruit individuals who are receiving outpatient services at the Minneapolis VA Medical Center, the University of Minnesota Department of Psychiatry, or the University of Minnesota Medical Center--Fairview. Patients will be referred by clinical staff from multiple departments including Mental Health, Polytrauma, and Social Work. Referral will be based on a clinical diagnosis of Schizophrenia or Schizoaffective disorder with medication refractory auditory hallucinations as assessed by the patient's clinical provider. Subjects will also have the ability to self-identify to flyers and local newspaper ads. Brunelin et al found a large and significant effect size (d=1.58, p<0.001) which the investigators have used to guide our power analysis. The investigators power analysis was performed for three arms using an alpha of 0.025, a power of 0.8, and a desired effect size of 1.00. This analysis results in a need for approximately 20 subjects per arm.

Pre-screening.

In order to reduce subject burden, the investigators will obtain a waiver of HIPAA authorization and informed consent for recruitment and screening to allow potential subjects to be pre-screened by chart review and in person or by telephone prior to scheduling potential participants for initial visit. Potential participants will be provided with information about the study and asked a series of questions to determine if they meet basic inclusion/exclusion criteria, such as a history of MRAH. They will be told about the basic aims of the study, and those interested in participating will be scheduled for an initial visit at which time they will complete consent paperwork.

Initiation Visit

The initiation visit (visit 1) starts with completion of informed consent, HIPAA, and the Modified Dysken Tool to assess capacity to consent. The participant must score 7 / 10 on the Dysken Tool in order to participate in the study. Should the participant score less than 7, s/he will be offered remedial teaching and re-assessment. Should the subject agree via consent and demonstrate capacity to consent, s/he is enrolled into the study. A full baseline evaluation is then performed. This includes assessment via MINI, MUPS, PANSS, AHRS, PSYRATS and Edinburgh Handedness Inventory.

Treatment Visits

Visits 2 - 10 are exclusively treatment visits. At each visit the participant completes the tES Side Effect Questionnaire (TSEQ) both pre and post treatment. Visits occur twice daily for 5 days. Visits must be spaced at least 2 hours apart. Depending on the arm participants have been randomized into, s/he will receive treatment with either tDCS, tRNS, or sham. Treatment will be provided using the Starstim Neurostimulator (Neuroelectrics, Inc.) This device has been approved for use in research in the United States without an investigational device exemption due to meeting criteria for non-significant risk. The same energetic parameters are used for both tDCS and tRNS (2mA for 20 min) as well as the same electrodes (SPONSTIM-25 25cm2 electrodes). Both tDCS and tRNS are initiated in a ramp-like fashion over 10s from 0mA to 2mA. Once at 2mA, tDCS is held constant for the entire session whereas the tRNS consists of an alternating current of 2mA with a 0mA offset applied at random frequencies over a range of 0.1 to 100 Hz. The sham procedure involves only 40 sec stimulation at 2mA and then drops to 0mA with 15msec pulses every 550msec. Should the participant not be able to tolerate a current of 2mA due to pain or irritation, the current will be decreased down to a minimum of 1.5mA. If 1.5 mA is still not tolerable, the participant will be removed from the study. Electrode placement is based on the international 10-20 electrode placement system. The anode is placed at the midpoint between F3 and FP1, a location corresponding approximately to the left dorsolateral prefrontal cortex, and the cathode placed at the midpoint between T3 and P3, a location corresponding to left temporo-parietal junction. Placement and parameters in tDCS are consistent with Brunelin et al, 2012). Placement and parameters in tRNS are consistent with. Stimulation setup and administration takes approximately 30 minutes.

Visit 11 is run the same as visits 2 - 10 but after completion of the final (10th) stimulation session, the subject will again complete the PANSS, AHRS, and PSYRATS. This visit typically takes 90 minutes.

Follow-Up Visits

Visits 12 - 14 are follow-up assessment only visits and occur at 1 month, 3 month, and 6 months post treatment. Participants will not receive stimulation but instead will be assessed via PANSS, AHRS, and PSYRATS.

Missed Visits

In the event that a participant misses a session of treatment, the session will be re-scheduled and treatment continued as soon as possible. The deviation from treatment will be noted in the study record.

Informed Consent Process

Consenting will take place in a private office at the Minneapolis VA Health Care System, University of Minnesota 717 Delaware office, the Ambulatory Research Center of the University of Minnesota Department of Psychiatry, or the UMPhysicians MINCEP clinic, depending on patient preference. Only the study staff obtaining consent, the subject, and any family members invited by the subject will be present. The research coordinator or other trained research staff will explain the study to the participants. After explaining the study, the participants will be allowed as much time as needed to review the HIPAA and consenting documents and ask any questions that might arise before making the decision to participate. If necessary, participants can delay participation for up to a week. Subjects will be allowed to review the consent form in private for as long as they need. Subjects will be allowed to ask any and all questions prior to providing consent. Study personnel obtaining consent will emphasize first and foremost that the study is voluntary and will not influence that subject's clinical care through the VA Medical Center, University of Minnesota Medical Center--Fairview, or the University of Minnesota Department of Psychiatry. To ensure comprehension of the information provided in the informed consent forms, participants will be asked to complete the Modified Dysken Tool and answer 7 out of 10 questions correctly.

Indications of Lack of Capacity to Consent

1. Potential participant has severe formal thought disorder that does not allow him or her to ask understandable questions or to answer the questions on the Dysken Tool
2. Potential participant is unable to maintain attention to the description of the consent form long enough to perceive the individual basic points in the consent form
3. Potential participant, either due to catatonia or otherwise, the potential participant cannot ask questions or respond sufficiently to indicate agreement
4. Potential participant expresses delusions related to the research protocol that significantly distort his or her basic understanding of the research.

No participant will be under legal commitment at the time of their consent or during their participation in the study.

Data Analysis

Data will be analyzed for group by time effects of stimulation method as compared to sham. Tolerability will also be assessed by looking at total side effect score compared to stimulation type. The data will be further analyzed using a clustering technique to understand the impact of symptom cluster and severity on overall treatment response.

Potential Risks and Benefits

This study involves the use of a tES device. With tES, both tDCS and tRNS are considered to be safe brain stimulation techniques that rarely result in adverse events. There is currently no evidence of serious side-effects. Criteria for discontinuation that may rarely occur are sores at the tCS administration site, headaches that impair global functioning, and worsening psychosis. Mild side-effects that typically resolve upon discontinuation tCS include light itching under the electrode at the beginning of administration, headache, fatigue, and nausea. The participant may choose to discontinue stimulation at any time during the session if experiencing discomfort or side effects. No other risks are anticipated. Nonetheless, in order to minimize risks, study staff will be using standards of administration that have been shown to be safe in numerous other studies and across more than 2000 studies using tES; this includes length of administration, magnitude of the current, size of electrode sponges used, and method of applying stimulation. Any unanticipated problems or adverse events will be reported according to MVAHCS standard operating procedure.

Study staff will use private (medical or educational) records during the recruitment process. Therefore, the use of protected health information may be associated with negative feelings about sharing medical/educational history. Participants may experience mild stress and/or discomfort with completing surveys/interview. Participants could also experience temporary feelings of stress or mental fatigue due to the behavioral assessment measures used in the study.

In addition, breach of confidentiality is a potential risk due to the use of sensitive private information. The results of this study may be published or presented but the participant's identity and records will not be revealed unless required by Federal Law. A Federal Law allows the U.S. Food and Drug Administration, Office for Human Research Protections, Government Accountability Office and other Federal agencies, the Research and Development Committee, representatives of USAMRMC, Henry M. Jackson Foundation, and/or the Institutional Review Board (IRB)/Human Studies Subcommittee of the VA Medical Center or University of Minnesota to review records. Because of the need for these inspections, absolute confidentiality cannot be guaranteed. However, every effort would be made to minimize these risks by providing the participant with a unique numerical identifier at the beginning of the study in order to protect their actual identification and maintain complete confidentiality.

It is possible that a participant may have a reduction of symptoms from the tES treatment but there are no anticipated direct or societal benefits to participation in this research project.

Research Monitor

A MVAHCS or University of Minnesota staff will act as an independent research monitor for this study. Her/His duties may include discussing the research protocol and recruitment with the investigator and staff, monitoring utilization of the tES device, follow-up with any participants in which an adverse event was reported, and reporting findings to the IRB.

Discontinuation Criteria

Sores at the tES administration site Headaches that impair global functioning Worsening psychosis

Privacy, Confidentiality, and Information Security

Self-report data will be collected on paper and scanned and stored in a password protected database behind the MVAMC or University of Minnesota firewalls. All personal identifiers will be stored on the consent form and in a master participant list within the database. All other documents will contain the unique participant ID. All paper documents related to this study will be stored in a locked file cabinet within locked research study offices. Access to research data and documents will be restricted to research personnel listed on the study protocol.

All data will be maintained at the MVAHCS and University of Minnesota indefinitely per requisite data retention policies. No data will be destroyed. Information regarding research results will not be shared with study participants.

ELIGIBILITY:
Inclusion Criteria

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder
* Age 18 to 64
* Experiencing medication refractory auditory hallucinations
* No antipsychotic medication changes or hospitalizations in the previous 4 weeks
* No substance dependence in the past six months and no substance abuse in the past month
* No clinically significant head injury or neurological disease
* Sufficient spoken English so as to be able to comprehend testing procedures
* No diagnosis of mental retardation or pervasive developmental disorder, i.e. premorbid IQ not less than 70
* Ability to give informed consent

Exclusion Criteria

* History of seizures or epilepsy
* History of metallic cranial plates, screws, or implanted device
* History of craniotomy
* History of eczema on the scalp
* Diagnosis of bipolar disorder
* Diagnosis of major depression with psychotic features
* Unable to give informed consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- 5775 Wayzata Blvd Suite 200, Saint Louis Park, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carter DM, Mackinnon A, Howard S, Zeegers T, Copolov DL. The development and reliability of the Mental Health Research Institute Unusual Perceptions Schedule (MUPS): an instrument to record auditory hallucinatory experience. Schizophr Res. 1995 Aug 1;16(2):157-65. doi: 10.1016/0920-9964(94)00069-k. PMID 7577769
- [Background] Nitsche MA, Doemkes S, Karakose T, Antal A, Liebetanz D, Lang N, Tergau F, Paulus W. Shaping the effects of transcranial direct current stimulation of the human motor cortex. J Neurophysiol. 2007 Apr;97(4):3109-17. doi: 10.1152/jn.01312.2006. Epub 2007 Jan 24. PMID 17251360
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- [Background] Hoffman RE, Hawkins KA, Gueorguieva R, Boutros NN, Rachid F, Carroll K, Krystal JH. Transcranial magnetic stimulation of left temporoparietal cortex and medication-resistant auditory hallucinations. Arch Gen Psychiatry. 2003 Jan;60(1):49-56. doi: 10.1001/archpsyc.60.1.49. PMID 12511172
- [Background] Lawrie SM, Buechel C, Whalley HC, Frith CD, Friston KJ, Johnstone EC. Reduced frontotemporal functional connectivity in schizophrenia associated with auditory hallucinations. Biol Psychiatry. 2002 Jun 15;51(12):1008-11. doi: 10.1016/s0006-3223(02)01316-1. PMID 12062886
- [Background] Slotema CW, Aleman A, Daskalakis ZJ, Sommer IE. Meta-analysis of repetitive transcranial magnetic stimulation in the treatment of auditory verbal hallucinations: update and effects after one month. Schizophr Res. 2012 Dec;142(1-3):40-5. doi: 10.1016/j.schres.2012.08.025. Epub 2012 Sep 30. PMID 23031191
- [Background] Vanneste S, Fregni F, De Ridder D. Head-to-Head Comparison of Transcranial Random Noise Stimulation, Transcranial AC Stimulation, and Transcranial DC Stimulation for Tinnitus. Front Psychiatry. 2013 Dec 18;4:158. doi: 10.3389/fpsyt.2013.00158. eCollection 2013. PMID 24391599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The PI for this study has left the institution. After extensive effort to locate more information, only limited study data is available. 3 participants were enrolled, however no baseline data was collected/is available.
Groups:
- Active tDCS: Current (2mA) is initiated in a ramp-like fashion over 10s from 0mA to 2mA using (SPONSTIM-25 25cm2 electrodes). The current is held constant for 20 min. Then the current is decreased in a ramp-like fashion over 10s from 2mA to 0mA.
  Transcranial Direct Current Stimulation: Energetic parameters are 2mA for 20 min with SPONSTIM-25 25cm2 electrodes. Current delivery is initiated in a ramp-like fashion over 10s from 0mA to 2mA.
- Active tRNS: Current (2mA) is initiated in a ramp-like fashion over 10s from 0mA to 2mA using (SPONSTIM-25 25cm2 electrodes). Once at 2mA, an alternating current of 2mA with a 0mA offset is applied at random frequencies over a range of 0.1 to 100 Hz. This is performed for 20 minutes. Then the current is decreased in a ramp-like fashion over 10s from 2mA to 0mA.
  Transcranial Random Noise Stimulation: Energetic parameters are 2mA for 20 min with SPONSTIM-25 25cm2 electrodes. Current delivery is initiated in a ramp-like fashion over 10s from 0mA to 2mA.
Period: Overall Study
Arm/Group | Sham | Active tDCS | Active tRNS
Started | 3 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 3 | 0 | 0
Not completed — Study Termination | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI for this study has left the institution. After extensive effort to locate more information, only limited study data is available. 3 participants were enrolled, however no baseline data was collected/is available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham | Active tDCS | Active tRNS | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Total Score of the Auditory Hallucinations Rating Scale
Time Frame: At 1 week and 1 month post treatment.
Population: as for baseline characteristics
Arm/Group | Sham | Active tDCS | Active tRNS
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Safety and Tolerability of Treatment Based on the Stimulation Side Effect Questionnaire
Time Frame: 1 week
Population: as for baseline characteristics
Arm/Group | Sham | Active tDCS | Active tRNS
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The PI for this study has left the institution. After extensive effort to locate more information, only limited study data is available. 3 participants were enrolled, however no data was collected/is available.
Description: The PI for this study has left the institution. After extensive effort to locate more information, only limited study data is available. 3 participants were enrolled, however no data was collected/is available. Treatment procedures were never initiated, therefore no participants were at risk of experiencing adverse events.
Arm/Group | Sham | Active tDCS | Active tRNS
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No